CLINICAL TRIAL: NCT01650558
Title: Randomized, Open-label Controlled Trial of Daily Trimethoprim-sulfamethoxazole or Weekly Chloroquine Among Adults on Anti-retroviral Therapy in Malawi
Brief Title: Daily Trimethoprim-sulfamethoxazole or Weekly Chloroquine Among Adults on ART in Malawi
Acronym: TSCQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Miriam Laufer, Associate Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HP-00043360; DAIDS ES-10822; U01AI089342-01A1 (NIH)
Record Dates: First submitted 2012-07-06; First posted 2012-07-26 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: HIV
Keywords: Malaria; HIV; Prophylaxis; Antiretroviral therapy
MeSH Terms: conditions — Malaria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care Prophylaxis (TS) (Active Comparator): Standard of care prophylaxis with daily trimethoprim sulfamethoxazole (TS).
  Interventions: Drug: Standard of Care prophylaxis
- Chloroquine (CQ) prophylaxis (Experimental): Discontinuation of standard of care TS prophylaxis and starting weekly chloroquine prophylaxis
  Interventions: Drug: Chloroquine (CQ) prophylaxis
- Discontinuation of standard of care (No Intervention): Control arm - Discontinuation of standard of care trimethoprim sulfamethoxazole.

INTERVENTIONS:
Drug: Standard of Care prophylaxis — Daily trimethoprim sulfamethoxazole
  Other Names: Bactrim; Co-trimoxazole
  Arms: Standard of Care Prophylaxis (TS)
Drug: Chloroquine (CQ) prophylaxis — Discontinue standard of care and start weekly CQ.
  Other Names: Aralen
  Arms: Chloroquine (CQ) prophylaxis

SUMMARY:
The purpose of this study is to determine if there is a benefit to taking trimethoprim-sulfamethoxazole (TS) as prophylaxis among HIV positive adults who have viral load suppression and a good clinical response on anti-retroviral therapy (ART). If there is a benefit, then is it due to antimalarial or antibacterial properties.

The investigators hypothesize that there will be a long-term benefit on survival and disease control in the context of prophylaxis and that the benefit will largely be attributed to prevention of malaria. The main study hypothesis is that 1)TS and chloroquine (CQ) will decrease the rates of morbidity and mortality among adults after 6 or more months of ART and 2) CQ prophylaxis will be associated with more prolonged viral suppression and higher CD4 cell counts than TS prophylaxis or no prophylaxis.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, phase III trial of standard of care TS prophylaxis and CQ prophylaxis compared to no prophylaxis in adults receiving ART. Adults who have been receiving ART for at least six months with a good clinical response and provide informed consent and fulfill the eligibility criteria will be randomized to one of three arms: (1) to continue standard of care trimethoprim-sulfamethoxazole (TS) prophylaxis, (2) discontinue standard of care TS prophylaxis and begin weekly CQ prophylaxis or (3) discontinue standard of care TS prophylaxis. Participants will be asked to return to the research clinic every four weeks for the first 24 weeks then every 12 weeks thereafter, and any time they are ill to facilitate both active and passive follow-up of the study endpoints. Participation will last for 32 to approximately 66 months. Participants who develop a WHO clinical stage 3 or 4 illness, experience a sustained decline in their CD4 count below 200 cells/mm3, or who experience ART failure will be placed on standard of care TS prophylaxis. Those with confirmed ART failure will be evaluated for second-line therapy according to the Malawi Ministry of Health guidelines.

The study population will include up to 1500 Malawian adults aged 18 years or older living with HIV in or near Blantyre or Zomba, Malawi, Central Africa who have been receiving antiretroviral therapy for at least 6 months with good clinical response to ART, have an undetectable HIV viral load and a CD4 count >250/mm3.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Documented HIV-1 infection
* Initiation of ART through a government-sponsored ART program at least six months prior
* Undetectable HIV viral load (< 400 copies/mL)
* CD4 count > 250/mm3
* TS prophylaxis prescribed for at least the previous 2 months
* Intention to remain in the study area until the end of the study period
* Informed consent from participant
* Female study volunteers of reproductive potential must have a negative urine pregnancy test performed within 20 days before randomization.
* Female study volunteers of reproductive potential who participate in sexual activity that could lead to pregnancy must use contraception (male or female condoms, diaphragm or cervical cap with spermicide, intrauterine device, or hormone-based contraceptive) while receiving their assigned study drug and for one month after stopping the medications.

Exclusion Criteria:

* Severe acute illness (defined as requiring hospitalization at the time of screening or other conditions such as laboratory abnormalities as determined by the investigators)
* Chronic treatment (requiring therapy for > 14 days) or secondary prophylaxis (for toxoplasmosis, Pneumocystis pneumonia, or tuberculosis for example) with any drug with antimalarial or antibacterial activity
* History of hypersensitivity to antifolate drugs or CQ
* Laboratory exclusion criteria
* Hemoglobin < 8.0 gm/dL
* Platelet count < 50,000/mm3
* Absolute granulocyte count < 500/mm3
* Serum alanine aminotransferase (ALT) concentration > 210 U/L for men, >160 U/L for women
* Serum creatinine concentration > 3.3mg/dl (291.7µmol/L) for men, and > 2.7mg/dl (238.7µmol/L) for women)
* History of visual field or retinal changes
* History of preexisting auditory damage
* History of porphyria
* History of psoriasis
* History of liver disease
* History of seizure disorder
* History of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of ECG and cardiac conduction abnormality or cardiomyopathy
* History of myopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1499 (Actual)
Dates: Start 2012-11; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam K Laufer, MD, MPH, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- Malawi (2):
  - Blantyre Malaria Project Research Clinic, Blantyre
  - Tisungane Clinic, Zomba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laurens MB, Mungwira RG, Nampota N, Nyirenda OM, Divala TH, Kanjala M, Mkandawire FA, Galileya LT, Nyangulu W, Mwinjiwa E, Downs M, Tillman A, Taylor TE, Mallewa J, Plowe CV, van Oosterhout JJ, Laufer MK. Revisiting Co-trimoxazole Prophylaxis for African Adults in the Era of Antiretroviral Therapy: A Randomized Controlled Clinical Trial. Clin Infect Dis. 2021 Sep 15;73(6):1058-1065. doi: 10.1093/cid/ciab252. PMID 33744963
- [Derived] Mungwira RG, Laurens MB, Nyangulu W, Divala TH, Nampota-Nkomba N, Buchwald AG, Nyirenda OM, Mwinjiwa E, Kanjala M, Galileya LT, Earland DE, Adams M, Plowe CV, Taylor TE, Mallewa J, van Oosterhout JJ, Laufer MK; TSCQ Study Team. High burden of malaria among Malawian adults on antiretroviral therapy after discontinuing prophylaxis. AIDS. 2022 Oct 1;36(12):1675-1682. doi: 10.1097/QAD.0000000000003317. Epub 2022 Jul 15. PMID 35848575
- [Derived] Laurens MB, Mungwira RG, Nyirenda OM, Divala TH, Kanjala M, Muwalo F, Mkandawire FA, Tsirizani L, Nyangulu W, Mwinjiwa E, Taylor TE, Mallewa J, Blackwelder WC, Plowe CV, Laufer MK, van Oosterhout JJ. TSCQ study: a randomized, controlled, open-label trial of daily trimethoprim-sulfamethoxazole or weekly chloroquine among adults on antiretroviral therapy in Malawi: study protocol for a randomized controlled trial. Trials. 2016 Jul 18;17(1):322. doi: 10.1186/s13063-016-1392-3. PMID 27431995

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis: Participants will continue standard of care daily TS prophylaxis (two tablets each of 80 mg trimethoprim and 400 mg sulfamethoxazole or one tablet each of 160 mg trimethoprim and 800 mg sulfamethoxazole).
- Chloroquine (CQ) Prophylaxis: Participants will discontinue standard of care trimethoprim sulfamethoxazol prophylaxis and start weekly CQ prophylaxis at 300 mg.
- Discontinuation of Standard of Care (Control Arm): Participants will discontinue standard of care trimethoprim sulfamethoxazol prophylaxis and receive no prophylaxis.
Period: Overall Study
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Started | 500 | 500 | 499
Completed | 417 | 408 | 424
Not Completed | 83 | 92 | 75
Not completed — Migration out of study area | 61 | 71 | 56
Not completed — Lost to Follow-up | 10 | 13 | 6
Not completed — Death | 10 | 6 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Non-compliant participant | 1 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm) | Total
Number analyzed (Participants) | 500 | 500 | 499 | 1499
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 494 | 496 | 480 | 1470
  >=65 years | 6 | 4 | 19 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9.7) | 38.7 (9.6) | 39.4 (10.1) | 39.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 374 | 386 | 1135
  Male | 125 | 126 | 113 | 364
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 500 | 500 | 499 | 1499
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 500 | 500 | 499 | 1499

OUTCOME MEASURES:

1. Primary Outcome: Severe Events
Description: Incidence of severe events (composite of death and WHO stage 3 and 4 illness)
Time Frame: 22-66 months
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Number analyzed (Participants) | 500 | 500 | 499
Events per 100 participant-years | 3.3 | 4.2 | 4.2
Statistical Analysis 1: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Discontinuation of Standard of Care (Control Arm); Test type: Non-Inferiority — Will assess performance of each experimental group relative to TS with a noninferiority margin for 1-HR of 0.35 to test the null (1-HR ≥ 0.35) and alternative (1-HR < 0.35) hypotheses. Each experimental group will be declared noninferior to TS if the upper bound of the 95% confidence interval of 1-HR is below 0.35. For ease of interpretation, the HRs have been recast with TS as the reference group, such that HRs greater than 1 indicate an increase in the experimental hazard rate relative to TS; p <= 0.05, Poisson — P-Value is not adjusted for multiple comparisons; Rate ratio confidence intervals and p-values were adjusted for overdispersion using the Pearson's chi-square scale; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.89 to 1.82]
Statistical Analysis 2: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Chloroquine (CQ) Prophylaxis; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Poisson — P-Value is not adjusted for multiple comparisons; Rate ratio confidence intervals and p-values were adjusted for overdispersion using the Pearson's chi-square scale; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.89 to 1.83]

2. Secondary Outcome: Number of Participants With at Least One Detectable HIV Viral Load
Description: Number of participants who ever have a detectable viral load (>400 copies/ml).
Time Frame: Throughout study participation, measured every six months (2-5.5 years).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Number analyzed (Participants) | 500 | 500 | 499
Participants | 24 | 36 | 33
Statistical Analysis 1: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Discontinuation of Standard of Care (Control Arm); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Fisher Exact — No adjustment for multiple comparisons was made; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.83 to 2.30]
Statistical Analysis 2: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Chloroquine (CQ) Prophylaxis; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Fisher Exact — No adjustment for multiple comparisons was made; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.91 to 2.49]

3. Secondary Outcome: CD4 Cell Count
Description: Number of Participants with at Least One CD4 Count <200
Time Frame: Every 6 months for 22-66 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Number analyzed (Participants) | 500 | 500 | 499
Participants | 24 | 23 | 27
Statistical Analysis 1: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Discontinuation of Standard of Care (Control Arm); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Fisher Exact — No adjustments for multiple comparisons were made; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.66 to 1.93]
Statistical Analysis 2: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Chloroquine (CQ) Prophylaxis; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Fisher Exact — No adjustments for multiple comparisons were made; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.55 to 1.68]

4. Secondary Outcome: WHO HIV Stage 2, 3, 4 Illness
Description: Incidence of any WHO HIV stage 2, 3, or 4 illness
Time Frame: 32-66 months
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Number analyzed (Participants) | 500 | 500 | 499
Events per 100 participant-years | 4.0 | 5.7 | 5.8
Statistical Analysis 1: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Discontinuation of Standard of Care (Control Arm); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Poisson — No adjustments for multiple comparisons were made; Rate ratio confidence intervals and p-values were adjusted for overdispersion using the Pearson's chi-square scale; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [1.07 to 2.00]
Statistical Analysis 2: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Chloroquine (CQ) Prophylaxis; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Poisson — No adjustments for multiple comparisons were made; Rate ratio confidence intervals and p-values were adjusted for overdispersion using the Pearson's chi-square scale; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [1.04 to 1.96]

5. Secondary Outcome: Bacterial Infections and Malaria
Description: Incidence of bacterial infections and malaria
Time Frame: 32-66 months
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Number analyzed (Participants) | 500 | 500 | 499
Events per 100 participant-years | 27.8 | 37.4 | 36.3
Statistical Analysis 1: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Discontinuation of Standard of Care (Control Arm); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Poisson — No adjustments for multiple comparisons were made; Rate ratio confidence intervals and p-values were adjusted for overdispersion using the Pearson's chi-square scale; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [1.11 to 1.55]
Statistical Analysis 2: Comparison: Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis vs Chloroquine (CQ) Prophylaxis; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p <= 0.05, Poisson — No adjustments for multiple comparisons were made; Rate ratio confidence intervals and p-values were adjusted for overdispersion using the Pearson's chi-square scale; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.14 to 1.58]

6. Secondary Outcome: Adverse Events Greater Than or Equal to Grade 3 That Are Related to the Study Product
Description: Occurrence of adverse events that are greater than or equal to Grade 3 that require discontinuation of TS or CQ prophylaxis
Time Frame: 32-66 months
Measure: Number; unit: Events per 100 participant-years
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazol (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
Number analyzed (Participants) | 500 | 500 | 499
Events per 100 participant-years | 0 | 0.24 | 0

7. Other Pre Specified Outcome: Bacterial or Malaria Infection With CQ or TS Resistant Organism
Description: Occurrence of bacterial or malaria infection with CQ or TS resistant organism
Time Frame: 32-66 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Clinical and Parasitological Response to Antimalarial Therapy
Description: Clinical and parasitological response to antimalarial therapy in cases of uncomplicated malaria
Time Frame: 32-66 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 to 5.5 years
Groups:
- Standard of Care Trimethoprim Sulfamethoxazo (TS) Prophylaxis: Participants will continue standard of care daily TS prophylaxis (two tablets each of 80 mg trimethoprim and 400 mg sulfamethoxazole or one tablet each of 160 mg trimethoprim and 800 mg sulfamethoxazole).
Arm/Group | Standard of Care Trimethoprim Sulfamethoxazo (TS) Prophylaxis | Chloroquine (CQ) Prophylaxis | Discontinuation of Standard of Care (Control Arm)
All-Cause Mortality (participants affected / at risk) | 10/500 | 6/500 | 8/499
Serious Adverse Events (participants affected / at risk) | 72/500 | 99/500 | 116/499
Other Adverse Events (participants affected / at risk) | 488/500 | 483/500 | 488/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Trimethoprim Sulfamethoxazo (TS) Prophylaxis (N=500) | Chloroquine (CQ) Prophylaxis (N=500) | Discontinuation of Standard of Care (Control Arm) (N=499)
Infections (Infections and infestations) | 22 (24) | 32 (36) | 40 (48)
Pregnancy, puerperium and perinatal (Pregnancy, puerperium and perinatal conditions) | 15 (21) | 26 (29) | 29 (32)
Nervous (Nervous system disorders) | 9 (9) | 11 (20) | 7 (8)
Injuries (Injury, poisoning and procedural complications) | 10 (10) | 7 (7) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 8 (8) | 8 (9)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 5 (5) | 9 (9)
Surgical and medical (Surgical and medical procedures) | 5 (5) | 6 (6) | 6 (6)
General (General disorders) | 2 (2) | 4 (6) | 6 (6)
Reproductive system (Reproductive system and breast disorders) | 3 (3) | 6 (7) | 3 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 3 (5)
Blood (Blood and lymphatic system disorders) | 4 (4) | 1 (2) | 2 (2)
Psychiatric (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2)
Eye (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Vascular (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Metabolism (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatobiliary (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Renal (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Trimethoprim Sulfamethoxazo (TS) Prophylaxis (N=500) | Chloroquine (CQ) Prophylaxis (N=500) | Discontinuation of Standard of Care (Control Arm) (N=499)
Infections (Infections and infestations) | 414 | 428 | 443
General (General disorders) | 304 | 267 | 312
Investigations (Investigations) | 298 | 307 | 278
Gastrointestinal (Gastrointestinal disorders) | 248 | 243 | 291
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 256 | 223 | 264
Blood (Blood and lymphatic system disorders) | 240 | 222 | 205
Nervous (Nervous system disorders) | 217 | 209 | 224
Skin (Skin and subcutaneous tissue disorders) | 140 | 133 | 138
Eye (Eye disorders) | 122 | 130 | 126
Reproductive system (Reproductive system and breast disorders) | 85 | 94 | 93
Injuries (Injury, poisoning and procedural complications) | 85 | 82 | 79
Respiratory (Respiratory, thoracic and mediastinal disorders) | 59 | 65 | 59
Vascular (Vascular disorders) | 17 | 29 | 31
Pregnancy, puerperium and perinatal (Pregnancy, puerperium and perinatal conditions) | 17 | 27 | 29
Metabolism (Metabolism and nutrition disorders) | 23 | 26 | 22
Ear and labyrinth (Ear and labyrinth disorders) | 18 | 24 | 18
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 23 | 16
Cardiac (Cardiac disorders) | 13 | 15 | 19
Renal (Renal and urinary disorders) | 11 | 17 | 19
Psychiatric (Psychiatric disorders) | 7 | 10 | 5
Surgical and medical (Surgical and medical procedures) | 6 | 6 | 7
Hepatobiliary (Hepatobiliary disorders) | 2 | 2 | 3
Endocrine (Endocrine disorders) | 1 | 1 | 2
Congenital, familial and genetic (Congenital, familial and genetic disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT01650558/Prot_SAP_000.pdf